## Association of Acupuncture and Cupping in Advanced Knee Osteoarthritis NCT 04168593

## Statistical analysis

The evaluation of the primary objective will be carried out by comparing the measures of the differences in the values between the initial and final WOMAC-Dor. To verify whether the median of the differences between the therapeutic groups showed a significant variation between the interventions, we used the non-parametric Kruskal-Wallis test adjusted for ties.

In assessing the amount of rescue pain medication used before and after treatment, we used the Chi Square test.

We used the concept of Intent to Treat (ITT) for statistical analysis purposes, that is, all recruited participants, even if they did not complete the proposed 10-session treatment, were included in the final analysis.

All the data were collected in the first interview and after 5 weeks treatment